CLINICAL TRIAL: NCT06293170
Title: Automated Screening for Clinically Ascertained Loss of Cerebral Functions in Patients With Severe Brain Damage - an Interventional Cluster Randomized Trial (DETECT-IVE)
Brief Title: Automated Screening for Clinically Ascertained Loss of Cerebral Functions
Acronym: DETECT-IVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Kristian Barlinn, Principal Investigator, Technische Universität Dresden
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Screening
Other Study IDs: 2024-DETECTIVENEUROLOGYUKD0001
Record Dates: First submitted 2024-02-21; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Irreversible Loss of Brain Function (ILBF)
Keywords: screening; detection; irreversible loss of brain function; death by neurologic criteria; brain death; organ donation
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Conventional care alone
  Interventions: Other: Conventional care
- DETECT (Experimental): DETECT in addition to conventional care will be initiated according to randomization plan
  Interventions: Other: DETECT; Other: Conventional care

INTERVENTIONS:
Other: DETECT — DETECT periodically processes real-time data from the corresponding electronic medical record system to screen for a combination of coma, indicated by a Richmond Agitation Sedation Scale (RASS) score of - 4 or - 5 or Glasgow Coma Scale (GCS) score of 6-3, along with manually assessed absence of bilateral pupillary light reflexes. Both findings are considered early indicators of impending ILBF. In case of positive screening results, an automated notification will be sent via the hospital's email server to the corresponding transplant coordinators and intensivists. The email sent aims to prompt clinical assessment of the reported patient and, if necessary, initiate a guideline-based ILBF examination.
  Arms: DETECT
Other: Conventional care — Conventional care

SUMMARY:
Rationale: The low organ donation rate in Germany is associated with the inadequate identification of patients at risk of developing irreversible loss of brain function (ILBF; i.e. brain death). An automated digital screening tool, DETECT (AutomateD ScrEening for Clinically AscerTainEd Loss of Cerebral FuncTions in Patients with Severe Brain Damage), has been developed to prospectively identify intensive care patients who are at risk of developing ILBF.

Objective: The objective of the study is to evaluate the effectiveness of an automated digital screening tool in the identification of patients with severe brain damage who are at risk of impending ILBF compared to standard practice without digital support.

Study design: Stepped-Wedge, multicenter, cluster-randomized, controlled trial

Study population: The study includes patients aged 18 years or older with primary and/or secondary acute brain damage, requiring mechanical ventilation, and who are deceased upon hospital discharge.

Intervention: DETECT periodically processes real-time data from the corresponding electronic medical record system to screen for a combination of coma, indicated by a Richmond Agitation Sedation Scale (RASS) score of - 4 or - 5 or Glasgow Coma Scale (GCS) score of 6-3, along with manually assessed absence of bilateral pupillary light reflexes. Both findings are considered early indicators of impending ILBF. In case of positive screening results, an automated notification will be sent via the hospital's email server to the corresponding transplant coordinators and intensivists. The email sent aims to prompt clinical assessment of the reported patient and, if necessary, initiate a guideline-based ILBF examination.

Primary study endpoint: The primary endpoint is the identification of patients who eventually develop ILBF during hospitalization.

Secondary study endpoints: Secondary outcomes encompass the missed identification of potential ILBF cases (as retrospectively classified) and the rate of deceased organ donations. Upon completion of the study, a survey will be conducted to investigate the stakeholders' experiences with DETECT.

ELIGIBILITY:
Inclusion Criteria:

* Primary and/or secondary acute brain damage
* At least 18 years or older
* Necessity of mechanical ventilation
* Deceased upon hospital discharge

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with diagnosis of ILBF | 30 months
  The primary outcome is defined as proportion of patients with an eventual diagnosis of ILBF in accordance with the guidelines of the German Medical Association during hospitalization.

SECONDARY OUTCOMES:
Number of patients who undergo deceased organ donation | 30 months
  The secondary outcome is defined as proportion of patients who undergo deceased organ donation.
Number of patients in whom diagnosis of ILBF was missed | 30 months
  The secondary outcome is defined as the failure to identify potential cases of ILBF. This outcome measure will be determined through retrospective evaluation of all deceased cases who were not diagnosed with ILBF during hospitalization. For this purpose, independent neurointensivists will review computed tomography and/or magnetic resonance imaging scans for findings indicative of critical intracranial pressure such as severe hypoxic cerebral edema, intracerebral hemorrhage with intraventricular extension or space-occupying hemispheric infarction, in addition to clinical information. The final decision regarding the potential development of ILBF will be based on consensus between two neurointensivists.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Barlinn, MD, Principal Investigator — Faculty of Medicine and University Hospital Carl Gustav Carus, Technische Universität Dresden, Fetscherstraße 74, 01307, Dresden, Germany
Locations (1):
- Faculty of Medicine and University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Germany

REFERENCES:
- [Background] Trabitzsch A, Pleul K, Barlinn K, Franz V, Dengl M, Gotze M, Guldner A, Eberlein-Gonska M, Albrecht DM, Hugo C. An Automated Electronic Screening Tool (DETECT) for the Detection of Potentially Irreversible Loss of Brain Function. Dtsch Arztebl Int. 2021 Oct 15;118(41):683-690. doi: 10.3238/arztebl.m2021.0307. PMID 34551858
- [Background] Schoene D, Freigang N, Trabitzsch A, Pleul K, Kaiser DPO, Roessler M, Winzer S, Hugo C, Gunther A, Puetz V, Barlinn K. Identification of patients at high risk for brain death using an automated digital screening tool: a prospective diagnostic accuracy study. J Neurol. 2023 Dec;270(12):5935-5944. doi: 10.1007/s00415-023-11938-1. Epub 2023 Aug 25. PMID 37626244
- [Derived] Schoene D, Roessler M, Pleul K, Hoehne S, Trabitzsch A, Barnett D, Guenzel A, Huttner HB, Sedlmayr M, Gunther A, Barlinn K; DETECT-IVE Investigators. Automated screening for clinically ascertained loss of cerebral functions in patients with severe brain injury-study protocol for a cluster-randomized interventional trial. Trials. 2025 Dec 11;27(1):39. doi: 10.1186/s13063-025-09354-z. PMID 41382177
- See also: Related Info — https://www.detect-iha.de/